CLINICAL TRIAL: NCT01889719
Title: Phase I Study to Evaluate the Safety/Immunogenicity of Boost Immunizations With MVA-CMDR in Healthy Volunteers Previously Immunized With Anti-DEC-205 Monoclonal Antibody Targeted HIV Gag p24 Vaccine Plus Poly-ICLC (RV 365 / WRAIR #2006)
Brief Title: A Phase I Study to Evaluate the Safety and Immunogenicity of Heterologous Boost Immunizations With MVA-CMDR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SSC-0803
Record Dates: First submitted 2013-06-20; First posted 2013-06-28 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: HIV
Keywords: HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccination with MVA-CMDR Group 1 (Experimental): Six to 27 subjects who previously received vaccination with DEC-205, will receive vaccination with MVA-CMDR
  Interventions: Biological: MVA-CMDR
- Vaccination with MVA-CMDR Group 2 (Active Comparator): Six to 27 subjects who previously did not receive vaccination with DEC-205, will receive vaccination with MVA-CMDR
  Interventions: Biological: MVA-CMDR

INTERVENTIONS:
Biological: MVA-CMDR — injections of MVA-CMDR vaccine

SUMMARY:
This trial will investigate whether immunizations with an MVA recombinant HIV vaccine are safe and whether they will boost immune responses generated by immunizations with a dendritic cell (DC) targeted protein vaccine, DCVax-001, plus poly ICLC in healthy HIV-uninfected volunteers.

DETAILED DESCRIPTION:
This trial will investigate whether immunizations with an MVA recombinant HIV vaccine are safe and whether they will boost immune responses generated by immunizations with a dendritic cell (DC) targeted protein vaccine, DCVax-001, plus poly ICLC in healthy HIV-uninfected volunteers. Investigators propose to assess the quality of immunity elicited by immunizations with MVA-CMDR only or by booster immunizations with MVA-CMDR in volunteers previously immunized with a DC-targeted HIV vaccine. This vaccination regimen can provide the proof-of-concept that DC targeted protein vaccines can prime strong immune responses and therefore be valuable in combination with other vaccine modalities against HIV or other diseases.

ELIGIBILITY:
Inclusion Criteria:

* Have completed protocol SSC-710 and received either DCVax-001 plus poly ICLC, poly ICLC only or sterile saline. If less than 6 volunteers who originally received placebo (poly ICLC only or sterile saline) under protocol SSC_710 are willing to participate and are found eligible to participate in this proposed study, new volunteers can be enrolled as long as they are eligible according to the remaining inclusion and exclusion criteria below.
* Healthy adult males and females, as assessed by a medical history, physical exam, ECG, and laboratory tests;
* Age of at least 18 years of age on the day of screening and no greater than 62 years at time of vaccination;
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study (screening plus 12 months);
* In the opinion of the principal investigator or designee, has understood the information provided. (Written informed consent needs to be given before any study-related procedures are performed);
* Amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit;
* Assessed by the clinic staff as being at "low risk" for HIV infection on the basis of sexual behaviors within the 12 months prior to enrollment defined as follows:
* Sexually abstinent OR
* Had two or fewer mutually monogamous relationships with partners believed to be HIV-uninfected and who did not use illicit drugs (illicit drug use or abuse that includes any injection drugs, methamphetamines (crystal meth), heroin, cocaine, including crack cocaine or chronic marijuana abuse) OR
* Had two or fewer partners believed to be HIV-uninfected and who did not use illicit drugs (as defined above) and with whom he/she regularly used condoms for vaginal and anal intercourse;
* If sexually active female, willing to use one effective method of contraception (combined oral contraceptive pill; injectable contraceptive; diaphragm; Intra Uterine Device (IUD); condoms; anatomical sterility in self or partner) at least until 3 months after last immunization. All female volunteers must be willing to undergo urine pregnancy tests at time points as indicated in the Schedule of Procedures.

Exclusion Criteria:

* Confirmed HIV-1 or HIV-2 infection
* Any clinically significant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids immunosuppressive anticancer, or other medications considered significant by the trial physician within the last 6 months
* Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, myopericarditis, grand-mal epilepsy, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation
* History of clinically significant eczema or chronic urticaria
* Any laboratory value outside of reference range, with the exception of any non-clinically significant Grade I elevations of liver function tests (AST, ALT, direct/total bilirubin), electrolytes (Na, K, Cl, CO2), CBC, urinalysis as determined by the Principal Investigator or his designee
* Baseline ECG with features that would interfere with interpretation of myo/pericarditis including significant repolarization abnormality, bundle branch block, and AV block
* Within the 12 months prior to enrollment, the volunteer has had excessive daily alcohol use or frequent binge drinking or chronic marijuana abuse or any other use of illicit drugs
* Within the 12 months prior to enrollment, the volunteer has a history of newly-acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), pelvic inflammatory disease (PID), mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, hepatitis B (surface antigen, HbsAg) or hepatitis C (HCV antibodies);
* If female, pregnant, planning a pregnancy during the 3-month follow up period after last immunization, or lactating
* Receipt of a live attenuated vaccine within 30 days or other vaccine within 14 days prior to study vaccination
* Prior use of medications for HIV PrEP
* Receipt of an investigational product (not vaccine-related) within the last 12 months. Receipt of a non-HIV experimental vaccine(s) within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For subjects who have received control/placebo in an experimental vaccine trial, or who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the investigators on a case-by-case basis.
* History of severe local or systemic reaction to vaccination defined as:
* Local: extensive, indurated redness and swelling involving most of the major circumference of the arm, not resolving within 72 hours;
* Systemic: fever > 39.5°C within 48 hours, anaphylaxis, bronchospasm, laryngeal edema, circulatory collapse, convulsions or encephalopathy within 72 hours
* History of immediate type hypersensitivity reaction to eggs or egg products
* Major psychiatric illness
* In the opinion of the investigator, unlikely to comply with protocol

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of MVA-CMDR vaccine | 16 weeks
  safety and tolerability of two intramuscular injections of MVA-CMDR vaccine candidate in healthy HIV-uninfected volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Schlesinger, MD, Principal Investigator — Rockefeller Univesrity
Locations (1):
- The Rockefeller University, New York, New York, United States